CLINICAL TRIAL: NCT04072198
Title: Phase II Study on NIVolumab in Combination With FOLFOXIRI/Bevacizumab in First Line Chemotherapy of Advanced COloRectal Cancer RASm/BRAFm Patients
Brief Title: Nivolumab Plus FOLFOXIRI/Bevacizumab in First Line Chemotherapy of Advanced Colorectal Cancer RASm/BRAFm Patients
Acronym: NIVACOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico Italiano di Ricerca Clinica (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOIRC-03-2018
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; Bevacizumab; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOXIRI/Bevacizumab + Nivolumab (Experimental): Bevacizumab 5 mg/m2 Nivolumab 240 mg Irinotecan 165 mg/m2 iv (max 8 cycles) Oxaliplatin + leucovorin 200 mg/m2 (max 8 cycles) Fluorouracil 3200 mg/m2 (max 8 cycles)
  Interventions: Drug: Nivolumab; Drug: Bevacizumab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: Leucovorin; Drug: fluoruracil

INTERVENTIONS:
Drug: Nivolumab — 240 mg every 2 weeks for 8 cycles followed by maintenance
Drug: Bevacizumab — 5 mg/kg every 2 weeks for 8 cycles followed by maintenance
Drug: Irinotecan — 165 mg/m2 every 2 weeks for 8 cycles
Drug: Oxaliplatin — 85 mg/m2 every 2 weeks for 8 cycles
Drug: Leucovorin — 200 mg/m2 every 2 weeks for 8 cycles
Drug: fluoruracil — 3200mg/m2 every 2 weeks for 8 cycles

SUMMARY:
This is a multicentric single arm, open label trial. In this study patients candidated to a first line of chemotherapy for metastatic colorectal cancer will be treated with 8 cycles of folfoxiri plus bevacizumab plus nivolumab followed by a maintenance with bevacizumab plus nivolumab.

Patients who do not progress during chemotherapy phase will receive bevacizumab plus nivolumab as maintenance therapy.

Patients will be treated until disease progression, unacceptable toxicity or patient/physician decision.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentric phase II trial in which patients with metastatic colorectal cancer RASm/BRAFm patients will receive nivolumab in combination with FOLFOXIRI/Bevacizumab as first line chemotherapy.

Study screening will take place within 28 days prior to initiation of study treatment. At screening, every patient must have local RAS/BRAF known status. A centralized review of RAS/BRAF status will be performed during the study.

Eligible patients will be enrolled and begin treatment with FOLFOXIRI/bevacizumab plus nivolumab every 2 weeks for 8 cycles followed by maintenance with bevacizumab plus nivolumab every 2 weeks until disease progression, unacceptable toxicity or patient/physician decision. Bevacizumab will be administered intravenously at dose of 5 mg/kg every 2 weeks. Nivolumab will be administered intravenously at flat dose of 240 mg every 2 weeks.

Folfoxiri will be administered as 165 mg/m2 intravenous infusion of irinotecan for 60 min, followed by an 85 mg/m2 intravenous infusion of oxaliplatin given concurrently with leucovorin at a dose of 200 mg/m2 for 120 min, followed by a 3200 mg/m2 continuous infusion of fluorouracil for 48 h.

During the study treatment period, patients will be followed for safety based on AE assessments including vital signs, physical findings and clinical laboratory test results.

In order to guarantee the safety of the patients, the enrolment will be stopped when the 10th patient will start treatment. An Independent Monitoring Committee will evaluate the safety data of these patients and will decide if the study should be completed, amended or closed.

Efficacy will be evaluated by the investigator according to RECIST v1.1 every 8 weeks during treatment and then every 3 months for 3 years.

During the study baseline tumor blocks will be centrally analysed to determinate inflammatory infiltrate, MSI/MSS and PD-L1 status. The biological characterization and Tumor Mutation Burden (TMB) will be also analysed centrally.

Following discontinuation of study treatment, safety assessments will be conducted 30 days after the last study drug administration or until initiation of other anti-cancer therapy (whichever occurs first). Thereafter, patients will be followed for disease progression (unless this has already occurred), SAEs, anticancer therapy and survival. Follow-up will continue for up to 3 years.

A blood sample will be collected for all patients at baseline, prior to cycle 5, at the end of chemotherapy and at disease progression.

Quality of life will be assessed at baseline, every 4 weeks during treatment and study discontinuation visit.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male or female of 18-75 years of age on day of signing informed consent.
3. Histologically confirmed diagnosis of colorectal cancer RAS/BRAF mutated.
4. Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease.
5. Patients suitable for first line chemotherapy.
6. Life expectancy > 3 months.
7. At least one site of measurable disease per RECIST criteria.
8. Performance status of 0-1 on the ECOG Performance Scale.
9. Adequate organ function
10. Availability at baseline of a representative formalin-fixed, paraffin-embedded (FFPE) diagnostic tumor specimen, as primary and/or metastatic tumor tissue block or as fifteen 5-micron unstained slides are allowed (the neoplastic cell content of each tumor sample will be assessed and in those cases with neoplastic cells <50% a macro-dissection of the specimen will be performed, if possible).
11. If DPD status is known it must be wild type. No restriction are applied if DPD status in unknown.
12. Women of childbearing potential must have a negative blood pregnancy test within 24 hr prior to the start of study drug. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive.
13. Subjects and their partners must be willing to avoid pregnancy during the trial and until 5 months for WOCBP (Women of Childbearing Potential) and 7 months for male subjects with female partners of WOCBP after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the investigator (barriers contraceptive measure or oral contraception).

Exclusion Criteria:

1. Prior chemotherapy, excluded patient treated in neo/adjuvant setting at least 12 months before diagnosis of metastatic disease.
2. Radiotherapy to any site within 4 weeks before the study.
3. Serious, non-healing wound, ulcer, or bone fracture.
4. Evidence of bleeding diathesis or coagulopathy.
5. Uncontrolled hypertension and prior history of hypertensive crisis or hypertensive encephalopathy.
6. Systemic corticosteroids within 2 weeks of the first dose of nivolumab.
7. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment.
8. Additional malignancy in the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
9. Active and untreated brain (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are not using steroids for at least 7 days prior to trial treatment.
10. Any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (> 10 mg daily prednisone equivalent) or immunosuppressive medications except for syndromes which would not be expected to recur in the absence of an external trigger.
11. Evidence of interstitial lung disease, active non-infectious pneumonitis, or a history of grade 3 or greater pneumonitis.
12. Active infection requiring systemic therapy.
13. History of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
14. Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection.
15. Live vaccine within 30 days prior to the first dose of trial treatment.
16. Chronic, daily treatment with high-dose aspirin (>325 mg/day).
17. Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment.
18. Any previous venous thromboembolism > NCI CTCAE Grade 3.
19. History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment.
20. Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes.
21. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study.
22. Presence of colic prosthesis or stent.
23. History of any severe hypersensitivity reactions to any monoclonal antibody.
24. Women of childbearing potential who are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
ORR | 36 months
  To demonstrate that adding nivolumab to standard colorectal first line chemotherapy improves the Overall Response Rate as determinated using RECIST 1.1 criteria

SECONDARY OUTCOMES:
Safety of combination | 36 months
  Safety assessments will include the incidence, nature, and severity of Adverse Events (AEs)
OS | 36 months
  Evaluate the efficacy in terms of overall survival (OS) defined as the time from start of study drug to the date of death from any cause
TTP | 36 months
  To evaluate the Time To Progression (TTP) defined as the time between the date of start of study drug and the first date of documented progression, based on investigator assessment (as per RECIST 1.1 criteria), or death due to any cause, whichever occurs first
Duration of response | 36 months
  To evaluate the duration of response defined as the time between the date of first evidence of response (SD/PR/CR) and the date of documented progression or death due to any cause, whichever occurs first
Quality of life with QLQ-C30 questionnaire | 36 months
  To evaluate the quality of life of patients determinated with questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carmine Pinto, MD, Principal Investigator — Gruppo Oncologico Italiano di Ricerca Clinica
Locations (8):
- Italy (8):
  - Istituto Ospedaliero Fondazione Poliambulanza, Brescia
  - Arnas Garibaldi, Catania
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Nazionale Tumori Fondazione G.Pascale, Napoli
  - Istituto Oncologico Veneto, Padua
  - AUSL/IRCCS di Reggio Emilia, Reggio Emilia
  - Policlinico Universitario Campus Bio-Medico, Roma
  - IRCCS - Casa Sollievo della Sofferenza, San Giovanni Rotondo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Damato A, Bergamo F, Antonuzzo L, Nasti G, Iachetta F, Romagnani A, Gervasi E, Larocca M, Pinto C. FOLFOXIRI/Bevacizumab Plus Nivolumab as First-Line Treatment in Metastatic Colorectal Cancer RAS/BRAF Mutated: Safety Run-In of Phase II NIVACOR Trial. Front Oncol. 2021 Dec 14;11:766500. doi: 10.3389/fonc.2021.766500. eCollection 2021. PMID 34970487
- [Derived] Damato A, Iachetta F, Antonuzzo L, Nasti G, Bergamo F, Bordonaro R, Maiello E, Zaniboni A, Tonini G, Romagnani A, Berselli A, Normanno N, Pinto C. Phase II study on first-line treatment of NIVolumab in combination with folfoxiri/bevacizumab in patients with Advanced COloRectal cancer RAS or BRAF mutated - NIVACOR trial (GOIRC-03-2018). BMC Cancer. 2020 Aug 31;20(1):822. doi: 10.1186/s12885-020-07268-4. PMID 32867715